CLINICAL TRIAL: NCT03605303
Title: Clinical Evaluation of Etafilcon A Contact Lenses Using a Novel Molding Process
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated due to the released lenses not representing what will be made commercially available and thus the objectives could not be met
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6270
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Results first posted 2019-07-24 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Refractive Error Correction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CONTROL- etafilcon A current molding (Active Comparator): 1-Day ACUVUE® MOIST
  Interventions: Device: Test/Control; Device: Control/Test
- TEST- etafilcon A novel molding (Experimental): Investigational Contact Lens
  Interventions: Device: Test/Control; Device: Control/Test

INTERVENTIONS:
Device: Test/Control — Subjects that are between the ages of 18-70 years old and habitual wearers of hydrogel daily disposable contact lenses will be randomly assigned to Test/Control sequence with a 7 to 9-day washout period in between treatments
Device: Control/Test — Subjects that are between the ages of 18-70 years old and habitual wearers of hydrogel daily disposable contact lenses will be randomly assigned to Control/Test sequence with a 7 to 9-day washout period in between treatments

SUMMARY:
This study is a multi-site, group sequential, adaptive, randomized, double-masked, 2×2 crossover design, 1-week dispensing study. Subjects will wear bilaterally both Test and Control lenses in a random order for 1-week each as a daily disposable modality with a wash-out period of 1 week between the wearing periods.

ELIGIBILITY:
Inclusion Criteria:

-Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Must be at least 18 and not more than 70 years of age (including 70) at the time of screening.
4. The subject must be a habitual and adapted wearer of hydrogel daily disposable brand contact lens in both eyes (at least 1 month of daily wear).
5. The subject must have normal eyes (i.e., no ocular medications or infections of any type).
6. The subject's required spherical contact lens prescription must be in the range of -1.00 to -4.50 D in each eye.
7. The subject's refractive cylinder must be < 0.75 D in each eye.
8. The subject must have best corrected visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any systemic disease, autoimmune disease, or use of medication that may interfere with contact lens wear.
3. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
4. Any ocular infection.
5. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
6. Monovision or multi-focal contact lens correction.
7. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
8. History of binocular vision abnormality or strabismus.
9. Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV, by self-report).
10. Suspicion of or recent history of alcohol or substance abuse.
11. History of serious mental illness.
12. History of seizures.
13. Employee of investigational clinic (e.g., Investigator, Coordinator, Technician).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Total Eye Care, PA, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: On July 06, 2018 Johnson & Johnson Vision terminated this study prematurely after lens testing revealed that the lens thickness in the mid-periphery of the lens were thinner than the lens design targets. As of this date only 3 subjects were enrolled at 1 site.
Groups:
- Test/Control: Subjects that were radnomized to wear the Test lens during the period and the Control lens during the second period. Both study lens was was to be worn bilaterally for a period of 1-week each.
- Control/Test: Subjects that were radnomized to wear the Control lens during the period and the Test lens during the second period. Both study lens was was to be worn bilaterally for a period of 1-week each.
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Study Terminated | 2 | 1
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Subjects: All subjects enrolled into th study
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 1
  White | 1
  Native Hawaiian or Other Pacfic Islander | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort Scores
Description: Subjective assessment of comfort will be performed using the Contact Lens User ExperienceTM (CLUE) questionnaire. CLUE is a validated patient reported outcomes (PRO) questionnaire used to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a US contact-lens wearing population between 18 and 65 years of age. CLUE composite scores are derived using Item Response Theory (IRT) and follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. A 5-point increase in an average CLUE score translates into 10% shift in the distribution of scores for the population of soft disposable contact lens wearers.
Time Frame: 1-Week Follow-up
Population: Study terminated early. No data was analyzed.
Groups:
- Test: subjects that were randomized to receive the Test lens in either period of the study.
- Control: All subject that were randomized to the Control lens during either period of the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Overall Vision Score
Description: Subjective assessment of vision will be performed using the Contact Lens User ExperienceTM (CLUE) questionnaire. CLUE is a validated patient reported outcomes (PRO) questionnaire used to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a US contact-lens wearing population between 18 and 65 years of age. CLUE composite scores are derived using Item Response Theory (IRT) and follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. A 5-point increase in an average CLUE score translates into 10% shift in the distribution of scores for the population of soft disposable contact lens wearers.
Time Frame: 1-Week Follow-up
Population: Study terminated early. No data was analyzed.
Arm/Group | Test | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approxmiately 3 days per subject.
Groups:
- Test: Subjects that wore the Test lens during any time throughout the duration of the study.
- Control: Subjects that wore the Control lens during any time throughout the duration of the study.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

LIMITATIONS AND CAVEATS:
This study was terminated after additional lens metrology testing revealed that the lens thickness of the contact lenses were thinner than the lens design targets. This reduction in thickness may have altered the handling of the contact lenses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT03605303/Prot_SAP_000.pdf